CLINICAL TRIAL: NCT01822444
Title: Exploratory Phase II Clinical Trial Comprising Biomarker Analysis of Oxaliplatin Plus Fluorouracil/Leucovorin (FOLFOX) in Combination With Bevacizumab (Bvz) in First Line Treatment of Metastatic Colorectal Cancer (CRC) Expressing Mutant K-ras - AC-ANGIOPREDICT
Brief Title: ANGIOPREDICT. ICORG 12-16, V3
Status: Completed | Type: Observational
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: ICORG 12-16
Record Dates: First submitted 2013-02-25; First posted 2013-04-02 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Advanced Colorectal Cancer
Keywords: Colorectal Cancer; Advanced Colorectal Cancer; Metastatic Colorectal Cancer; Locally Advanced Colorectal Cancer; Colon Cancer; Rectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Intent-to-treat population with aCRC or mCRC: Advanced Colorectal Cancer with planned treatment with a aCRC or mCRC and who fulfil all inclusion and exclusion criteria
  Interventions: Other: Biomarker analysis

INTERVENTIONS:
Other: Biomarker analysis

SUMMARY:
Primary Objective:

The primary objective is to validate previously identified predictive/prognostic genomic DNA and expression biomarkers of response to combination bvz treatments in K-ras mutant advanced CRC (a CRC) or metastatic CRC (mCRC).

Secondary Objective:

1. To test the efficacy of bvz in combination with FOLFOX in patients with newly diagnosed advanced or metastatic K-ras mutant CRC and
2. To determine the progression free and overall survival of patients under first line FOLFOX + bvz in aCRC or mCRC.

DETAILED DESCRIPTION:
Study Design:

Type of Study: Exploratory, translational, multicenter and multinational Phase II study.

Patient Population:All patients from the intent-to-treat population with aCRC or mCRC, (incurable with any conventional multimodality approach) and who fulfil all inclusion and exclusion criteria.

Number of Patients: 224

Sample Type:

Serial tissue and blood samples will be collected before (week 0), during (week 6, month 3 and 6) and at the end of treatment (month 12).

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age.
2. Patients diagnosed with recurrent or de novo, locally advanced (unresectable) or metastatic adenocarcinoma of the colon or rectum.
3. Planned combination bevacizumab (bvz) treatment with either:

   * leucovorin, fluorouracil and oxaliplatin (FOLFOX)
   * capecitabine and oxaliplatin (XELOX)
   * leucovorin, fluorouracil and irinotecan (FOLFIRI)
   * capecitabine and irinotecan (XELIRI)
4. Naive for bvz
5. An evaluable site of disease
6. ECOG Performance status 0, 1, or 2
7. Adequate renal function as shown by serum creatinine ≤ 1.5 x ULN or GFR ≥ 50ml/min
8. Adequate hematopoietic function [white blood cell (WBC) count ≥ 3000/μl, absolute neutrophil count (ANC) ≥1500/μl, platelets ≥100 000/μl, haemoglobin level ≥ 9.0 g/dl]
9. Adequate end organ function, defined as the following: total bilirubin < 1.5 x ULN, SGOT and SGPT < 3.0 x ULN (in case of liver metastases SGOT and SGPT < 5.0 x ULN)
10. Ability to give signed informed consent prior to any screening procedures
11. FFPE Tissue is available

Exclusion Criteria:

1. Patient has received any other investigational product within 28 days of first day of study drug dosing
2. Patients having familial and/or hereditary CRC
3. CRC associated with ulcerative colitis
4. Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients from the intent-to-treat population with aCRC or mCRC, (incurable with any conventional multimodality approach) and who fulfil all inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Identification of biomarkers | 4 years
  Identification of biomarkers, which are predictive for response and/or prolonged PFS to FOLFOX/bvz combination therapy in aCRC or mCRC patients.

SECONDARY OUTCOMES:
Validation of identified biomarkers | 4 years
  Validation of identified biomarkers with regard to response rate/failure to further treatment strategy, PFS, overall survival (OS) and toxicity.

CONTACTS AND LOCATIONS:
Locations (17):
- Germany (8):
  - Private Practice Oncology, Speyer, Rhineland-Palatinate
  - Medizinische Klinik III, Universitaetsklinikum, Aachen
  - Onkologisches Zentrum, Deggendorf
  - University Hospital Saarland, Homburg
  - Gemeinschaftspraxis Haematologie/Onkologie, Lebach
  - Kilnikum Ludwigsburg, Ludwigsburg
  - Medizinische Klinik and Poliklinik Mainz, Mainz
  - Univeritaetsmedizin Mannheim, Mannheim
- Ireland (9):
  - Bon Secours Hospital, Cork
  - Cork University Hospital, Cork
  - St Vincent's University Hospital, Dublin
  - Beaumont Hospital, Dublin
  - St James Hospital, Dublin
  - The Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital, Dublin
  - Galway University Hospital, Galway
  - Sligo General Hospital, Sligo
  - Waterford Regional Hospital, Waterford

IPD SHARING:
Plan to Share IPD: Undecided